CLINICAL TRIAL: NCT00106938
Title: Carotid Angioplasty and Stenting Versus Endarterectomy in Asymptomatic Subjects Who Are at Standard Risk for Carotid Endarterectomy With Significant Extracranial Carotid Stenotic Disease (ACT I)
Acronym: ACT I
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Business decision and not a result of any patient or product safety issues.
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AVD-640-0052
Record Dates: First submitted 2005-04-01; First posted 2005-04-04 (Estimated); Results first posted 2014-10-21 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-06

CONDITIONS: Carotid Artery Disease; Carotid Stenosis; Stroke; Atherosclerosis
Keywords: Carotid stenting; Carotid endarterectomy; Carotid artery disease with severe narrowing of the artery; Stroke prevention
MeSH Terms: conditions — Carotid Artery Diseases; Carotid Stenosis; Stroke; Atherosclerosis | interventions — Methods; Endarterectomy, Carotid; Surgical Procedures, Operative

ARMS (2):
- 1 (Active Comparator): CAS group: 3:1 ratio of Carotid Artery Stenting (CAS) versus Carotid Endarterectomy (CEA).
  Subjects will be followed at 30 days, six (6), and 12 months post-procedure, and annually for four (4) additional years.
  Interventions: Device: Carotid artery stenting with filter (interventional)
- 2 (Active Comparator): CEA group: 3:1 ratio of Carotid Artery Stenting (CAS) versus Carotid Endarterectomy (CEA).
  Subjects will be followed at 30 days, six (6), and 12 months post-procedure, and annually for four (4) additional years.
  Interventions: Procedure: Carotid artery endarterectomy (surgical)

INTERVENTIONS:
Device: Carotid artery stenting with filter (interventional) — Carotid artery stenting with filter (interventional)
  Arms: 1
Procedure: Carotid artery endarterectomy (surgical) — Carotid artery endarterectomy (surgical)
  Arms: 2

SUMMARY:
The study is being conducted to demonstrate the non-inferiority of carotid artery stenting (CAS) using the Emboshield® Embolic Protection System with the Xact® Carotid Stent System to carotid endarterectomy (CEA) for the treatment of asymptomatic extracranial carotid atherosclerotic disease.

DETAILED DESCRIPTION:
Randomization for ACT 1 employs a 3:1 ratio of CAS versus CEA. A lead-in phase of up to 400 carotid stent subjects will provide investigators experience with the study devices prior to pivotal enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must be > 18 and < 80 years of age.
2. Female subjects of child bearing potential must have a documented negative pregnancy test within 30 days prior to the study procedure.
3. Subject must be asymptomatic, defined as no stroke or Transient Ischemic Attack [(TIA);(hemispheric or ocular)] within the 180 days prior to the procedure. Subjects who have experienced these neurological symptoms prior to the 180 day pre-procedure window will be eligible for enrollment. An independent study neurologist or independent study neurosurgeon must confirm the subject's neurological status.
4. Subjects taking warfarin may be included if their dosage is reduced before the procedure to result in an International Normalized Ratio (INR) of 1.5 or less. Warfarin may be restarted after the procedure.
5. The subject must sign a written informed consent prior to the procedure, using a form that is approved by the local institutional review board (IRB).
6. The subject must agree to return for all required follow-up visits.
7. Subject has a discrete lesion located in the internal carotid artery (ICA); the contiguous common carotid artery (CCA) may be involved.
8. Carotid stenosis ≥ 70% and ≤ 99% by carotid ultrasound or ≥ 70% and ≤ 99% stenosis (visual estimate) by angiography, without significant (> 60% by ultrasound or angiography) ICA/CCA contralateral stenosis.
9. Target ICA vessel diameter must be visually estimated to be:

   > 2.5 mm and < 7.0 for the Emboshield Pro or for the Emboshield NAV6, > 2.8 mm and < 6.2 for the Emboshield Gen 3 And > 4.0 mm and < 9.0 mm for the Xact stent treatment segment. An untreated contralateral ICA may be used for visual estimation when a highly stenosed lesion makes measurement of the target vessel inaccurate.
10. Based on the subject's anatomy, the Investigator should expect to successfully deliver the stent to the target lesion (absence of extreme tortuosity, etc.).
11. De novo target lesion that can be treated with a single stent.

Exclusion Criteria:

Each potential subject must be screened to ensure that they do not meet any of the following exclusion criteria. This screening is to be based on known medical history and data available at the time of eligibility determination and enrollment.

1. Subject is symptomatic and has had a stroke or exhibited TIA (hemispheric or ocular) within 180 days prior to randomization, which has been confirmed by an independent study neurologist or independent study neurosurgeon.
2. Subject is participating in another drug or device trial (IND or IDE) that has not completed the primary endpoint or that may potentially confound the results of this trial. Subject may be enrolled only once in this trial and may not participate in any other clinical trial during a 1-year period post-index procedure.
3. Subject has inability to understand and cooperate with study procedures or provide informed consent.
4. Subject has had an intracranial hemorrhage or hemorrhagic stroke within 1-year prior the index procedure.
5. Subject has dementia or has a neurological illness that may confound the neurological evaluation.
6. Subject has had a known untoward reaction to anesthesia or contrast media not able to be overcome by pre-treatment with medications.
7. Subject has history of intolerance or allergic reaction to any of the study medications including aspirin, Clopidogrel bisulfate (Plavix®) or Ticlopidine (Ticlid®), heparin or Bivalirudin (Angiomax™). Subjects must be able to tolerate a combination of aspirin and Clopidogrel/Ticlopidine.
8. Subject has Hemoglobin (Hgb) less than 10 gm/dL, platelet count <100,000/mm3 or >500,000/mm3, or known heparin associated thrombocytopenia.
9. Subject has an active bleeding diathesis or coagulopathy, or will refuse blood transfusions.
10. Subject has had a GI bleed that would interfere with antiplatelet therapy.
11. Subject has known cardiac sources of emboli, including paroxysmal or sustained atrial fibrillation (treated or untreated).
12. Subject has had an myocardial infarction (MI) within the previous 30 days.
13. Subject has any condition that limits their anticipated survival to less than 3 years.
14. Subject is a high risk surgical candidate defined as the presence of any one or more of a following medical conditions:

    1. Two or more proximal diseased coronary arteries of > 70% stenosis that have not or cannot be revascularized or < 30 days since revascularization.
    2. Ejection fraction < 30% or New York Heart Association (NYHA) heart failure functional class 3 or higher.
    3. Unstable angina, defined as angina at rest with ECG changes.
    4. On a list for major organ transplant or is being evaluated for such.
    5. Known history of respiratory insufficiency, forced expiratory volume (FEV1) < 30% (predicted).
    6. Chronic renal insufficiency (serum creatinine >2.5 mg/dL).
    7. Uncontrolled diabetes defined as fasting glucose > 400 mg/dL.
    8. Concurrent requirement for any invasive procedure 30 days pre- or post-procedure.
    9. Age ≥ 80 years.
15. Subject may be considered a non-surgical candidate for CEA as a result of one or more anatomic conditions or features which preclude normal surgical access or a high surgical risk because of the presence of any one or more anatomic conditions that present an increased potential for adverse events. These subjects are not eligible for enrollment.

    1. Subject has had radiation treatment to the neck.
    2. Subject has had a radical neck dissection.
    3. Surgically inaccessible lesions (i.e., lesions extending above the level of C2).
    4. Spinal immobility - inability to flex neck beyond neutral or kyphotic deformity.
    5. Presence of carotid artery dissection, aneurysm, pseudoaneurysm, arteritis or fibromuscular dysplasia (FMD) in the target vessel.
    6. Hemodynamically significant (>60%) stenosis of the right or left common carotid artery (LCCA/RCCA) below the clavicle.
    7. Presence of tracheostomy stoma.
    8. Contralateral laryngeal nerve paralysis.
    9. Previous carotid endarterectomy, extracranial-intracranial or carotid subclavian bypass procedure ipsilateral to the carotid stenosis.
    10. Severe hypertension (defined as blood pressure > Systolic of 180 mm Hg and/or a diastolic of 110 mm Hg) not adequately controlled by anti-hypertensive therapy at the time of study entry.
16. Severe vascular disease including tortuosity and/or occlusive disease that would preclude the safe introduction of a guiding catheter/sheath, cerebral protection device, balloon catheter, stent delivery system or stent placement. Severe tortuosity is defined as 2 or more >90 degree bend points within 3cm of the target stenosis. One of these bends will be considered to be present if the ICA branches from the CCA at a 90 degree angle. This includes aortic arch anatomy that is unacceptable for carotid stent placement.
17. Intraluminal filling defect thought to represent thrombus.
18. Excessive calcification: defined as fluoroscopic evidence of calcium that extends circumferentially around the target lesion and includes the majority of the atherosclerotic plaque.
19. Occlusion (TIMI 0 flow), or string sign of the ipsilateral common or internal carotid artery.
20. The target lesion requires treatment with a device other than percutaneous transluminal angioplasty (PTA) prior to stent placement.
21. Significant (> 60%) stenosis proximal or distal to the target lesion that might require revascularization or impede run off.
22. Presence of a previously placed intravascular stent in the ipsilateral carotid distribution.
23. Cerebral aneurysm (symptomatic or > 10 mm) or arteriovenous malformation (AVM) of the cerebral vasculature.
24. Bilateral carotid stenosis (ICA/CCA contralateral stenosis > 60% by ultrasound or angiography).

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1663 (Actual)
Dates: Start 2005-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon Matsumura, MD, Principal Investigator — University of Wisconsin, Madison; Kenneth Rosenfield, MD, Principal Investigator — Massachusetts General Hospital
Locations (62):
- United States (62):
  - St. Luke's Hospital-Phoenix, Phoenix, Arizona
  - Mayo Clinic, Phoenix, Arizona
  - Fogarty Clinical Research Inc./El Camino Hospital, Mountain View, California
  - Hoag Memorial Hospital, Newport Beach, California
  - St. Joseph Hospital, Orange, California
  - Kaiser Foundation Hospital-San Diego, San Diego, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Baptist Cardiac and Vascular Institute, Miami, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Hawaii Permanente Medical Group - Kaiser, Honolulu, Hawaii
  - Northwestern University Memorial Hospital, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - St. John's Hospital and Memorial Medical Center/ Prairie Heart Cooperative, Springfield, Illinois
  - Parkview Hospital, Fort Wayne, Indiana
  - Central Baptist Hospital, Lexington, Kentucky
  - University of Louisville, Louisville, Kentucky
  - Cardiovascular Institute of the South, Lafayette, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Harper University Hospital/Detroit Medical Center, Detroit, Michigan
  - McLaren Regional Medical Center, Flint, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - St. John's Mercy Medical Center, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Our Lady of Lourdes Medical Center, Camden, New Jersey
  - Albany Medical Center, Albany, New York
  - Millard Fillmore Hospital, Buffalo, New York
  - NYU Medical Center, New York, New York
  - Columbia Presbyterian Hospital, New York, New York
  - Lenox Hill Hospital, New York, New York
  - University of Rochester-Strong Memorial Hospital, Rochester, New York
  - St. Francis Hospital, Roslyn, New York
  - Duke University Medical Center, Durham, North Carolina
  - WakeMed Health and Hospital, Raleigh, North Carolina
  - Forsyth Medical Center, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Oregon Health and Science University Stroke Center, Portland, Oregon
  - Heritage Valley Health System, Beaver, Pennsylvania
  - Harrisburg Hospital / Pinnacle Health, Harrisburg, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center (UPMC), Pittsburgh, Pennsylvania
  - University of Pittsburgh Physicians Division of Vascular Surgery/Shadyside Medical, Pittsburgh, Pennsylvania
  - Allegheny General Hospital, Washington, Pennsylvania
  - St. Joseph's Medical Center/Berks Cardiologists, Wyomissing, Pennsylvania
  - Providence Hospital-SC, Columbia, South Carolina
  - North Central Heart Institute, Sioux Falls, South Dakota
  - The Stern Cardiovascular Center/Methodist Germantown Hospital, Germantown, Tennessee
  - Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - Mercy Medical West/Turkey Creek Medical Center, Knoxville, Tennessee
  - Westlake Medical Center/Seton Heart Institute, Austin, Texas
  - Heart Hospital of Austin, Austin, Texas
  - Dallas Veteran's Administration Medical Center, Dallas, Texas
  - Presbyterian Hospital of Dallas, Dallas, Texas
  - St. Luke's Episcopal Hospital, Houston, Texas
  - Chesapeake General Hospital/Sentara Norfolk General Hospital, Norfolk, Virginia
  - St. Mary's Hospital / Virginia Cardiovascular Specilists, Richmond, Virginia
  - Deaconess Medical Center, Spokane, Washington
  - University of Wisconsin, Madison, Wisconsin
  - St. Luke's Medical Center - Milwaukee, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Weinberg I, Beckman JA, Matsumura JS, Rosenfield K, Ansel GM, Chaturvedi S, Gray W, Metzger DC, Riles T, Shu Y, Wechsler L, Jaff MR. Carotid Stent Fractures Are Not Associated With Adverse Events: Results From the ACT-1 Multicenter Randomized Trial (Carotid Angioplasty and Stenting Versus Endarterectomy in Asymptomatic Subjects Who Are at Standard Risk for Carotid Endarterectomy With Significant Extracranial Carotid Stenotic Disease). Circulation. 2018 Jan 2;137(1):49-56. doi: 10.1161/CIRCULATIONAHA.117.030030. Epub 2017 Oct 5. PMID 28982691
- [Derived] Rosenfield K, Matsumura JS, Chaturvedi S, Riles T, Ansel GM, Metzger DC, Wechsler L, Jaff MR, Gray W; ACT I Investigators. Randomized Trial of Stent versus Surgery for Asymptomatic Carotid Stenosis. N Engl J Med. 2016 Mar 17;374(11):1011-20. doi: 10.1056/NEJMoa1515706. Epub 2016 Feb 17. PMID 26886419

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Asymptomatic subjects with extracranial internal carotid stenosis which was ≥70% & ≤99% by duplex ultrasound or ≥70% & ≤99% by angiography (visual estimate) with or without involvement of the contiguous common carotid artery, who could undergo carotid artery stenting/carotid endarterectomy and all follow-ups, were recruited starting from April 2005
Pre-assignment Details: 1453 patients were randomized to support the primary analysis; an additional 210 lead-in subjects were enrolled to allow investigators to gain experience with the study devices prior to randomizing subjects and were not part of the primary analysis.
Groups:
- CAS Group: CAS group: 3:1 ratio of Carotid Artery Stenting (CAS) versus Carotid Endarterectomy (CEA).
  Subjects will be followed at 30 days, six (6), and 12 months post-procedure, and annually for four (4) additional years.
- CEA Group: CEA group: 3:1 ratio of Carotid Artery Stenting (CAS) versus Carotid Endarterectomy (CEA).
  Subjects will be followed at 30 days, six (6), and 12 months post-procedure, and annually for four (4) additional years.
Period: Overall Study
Arm/Group | CAS Group | CEA Group
Started | 1089 | 364
Completed | 913 | 293
Not Completed | 176 | 71

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CAS Group | CEA Group | Total
Number analyzed (Participants) | 1089 | 364 | 1453
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 325 | 103 | 428
  >=65 years | 764 | 261 | 1025
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.7 (7.0) | 67.9 (6.9) | 67.7 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 423 | 157 | 580
  Male | 666 | 207 | 873
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 985 | 327 | 1312
  Hispanic or Latino | 38 | 12 | 50
  Pacific Islander | 0 | 1 | 1
  Black or African American | 45 | 16 | 61
  American Indian or Alaska | 1 | 0 | 1
  Asian | 10 | 4 | 14
  Other | 10 | 4 | 14
Region of Enrollment [Number; unit: participants]
  United States | 1089 | 364 | 1453

OUTCOME MEASURES:

1. Primary Outcome: Composite of Death, Stroke (Ipsilateral or Contralateral; Major or Minor) and Myocardial Infarction (DSMI) Through 30 Days Post-procedure, Plus Ipsilateral Stroke 31 to 365 Days.
Time Frame: 0 to 365 days
Measure: Number; unit: percentage of participants
Arm/Group | CAS Group | CEA Group
Number analyzed (Participants) | 1089 | 364
percentage of participants | 3.8 | 3.4

2. Secondary Outcome: Acute Device Success: Xact Carotid Stent
Description: Defined as attainment of final residual diameter stenosis of < 50% by Qualitative Comparative Analysis (QCA) (if QCA is not available, the visual estimate of diameter stenosis will be used) covering an area no longer than the original lesion with the study stent. (Routine post-dilatation of the stent may be included in this definition). Placement of an additional stent to treat a dissection or procedural complication as a bailout will not be considered a device success.
Time Frame: On day 0 after index procedure
Population: Device success is per device basis including the attempted devices only, including the attempted Carotid Artery Stenting (CAS) device only.
Measure: Number (95% Confidence Interval); unit: percentage of devices
Units Other Than Participants: devices
Arm/Group | CAS Group
Number analyzed (Participants) | 1025
Number analyzed (devices) | 1049
percentage of devices | 96.9 [95.6 to 97.8]

3. Secondary Outcome: Acute Device Success: Embolic Protection Device System
Description: Defined as successful deployment and retrieval of the filter in the absence of angiographic distal embolization.
Time Frame: On day 0 after index procedure
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Percentage of devices
Units Other Than Participants: Devices
Arm/Group | CAS Group
Number analyzed (Participants) | 1022
Number analyzed (Devices) | 1045
Percentage of devices | 97.8 [96.7 to 98.6]

4. Secondary Outcome: Procedural Success
Description: Procedural success is defined as the attainment of target lesion final residual diameter stenosis of < 50% by QCA (if QCA is not available, the visual estimate of diameter stenosis will be used) using any procedural method and freedom of Major Adverse Event at 30 days.
Time Frame: 0 to 30 days post procedure
Population: The analysis population is Procedure success is per subject basis including the attempted CAS (carotid artery stenting) procedure only. CEA group is not part of analysis population for procedure success.
Measure: Number; unit: percentage of participants
Arm/Group | CAS Group
Number analyzed (Participants) | 1025
percentage of participants | 95.6

5. Secondary Outcome: Composite Morbidity Measure
Description: A pre-specified composite Morbidity Measure (CMM) of cranial and peripheral nerve injury, vascular injury, non-cerebral bleeding, wound complications related to the neck incision or femoral puncture site, and other complications (anesthetic) at 30 days post-procedure.
Time Frame: 0 to 30 Days Post-procedure
Population: Intent-to-Treat (ITT) population
Measure: Number; unit: participants
Arm/Group | CAS Group | CEA Group
Number analyzed (Participants) | 1089 | 364
participants
  Composite morbidity measure | 31 | 17
  Cranial nerve injury | 1 | 4
  Peripheral nerve injury | 0.0 | 0.0
  Vascular injury | 8 | 3
  Non-cerebral bleeding | 21 | 6
  CEA wound or access artery wound | 3 | 4
  Other complications | 0 | 0

6. Secondary Outcome: Freedom From Clinically Indicated Target Lesion Revascularization(CI-TLR)
Description: Freedom from CI-TLR was defined as freedom from reintervention for ≥ 50% restenosis in recently symptomatic patients and ≥ 80% restenosis in asymptomatic patients.
Time Frame: 0 to 180 days
Measure: Number; unit: percentage of partcipants
Arm/Group | CAS Group | CEA Group
Number analyzed (Participants) | 1089 | 364
percentage of partcipants | 99.8 | 99.7

7. Secondary Outcome: Freedom From Clinically Indicated Target Lesion Revascularization
Description: Freedom from CITLR was defined as freedom from reintervention for ≥ 50% restenosis in recently symptomatic patients and ≥ 80% restenosis in asymptomatic patients.
Time Frame: 0 to 365 days
Measure: Number; unit: percentage of partcipants
Arm/Group | CAS Group | CEA Group
Number analyzed (Participants) | 1089 | 364
percentage of partcipants | 99.4 | 97.4

8. Secondary Outcome: Freedom From Clinically Indicated Target Lesion Revascularization
Description: as for outcome 7
Time Frame: 0 to 730 days
Measure: Number; unit: percentage of partcipants
Arm/Group | CAS Group | CEA Group
Number analyzed (Participants) | 1089 | 364
percentage of partcipants | 98.7 | 96.7

9. Secondary Outcome: Freedom From Clinically Indicated Target Lesion Revascularization
Description: as for outcome 7
Time Frame: 0 to 1095 days
Measure: Number; unit: percentage of partcipants
Arm/Group | CAS Group | CEA Group
Number analyzed (Participants) | 1089 | 364
percentage of partcipants | 98.4 | 96.7

10. Secondary Outcome: Freedom From Clinically Indicated Target Lesion Revascularization
Description: as for outcome 7
Time Frame: 0 to 1460 days
Measure: Number; unit: percentage of partcipants
Arm/Group | CAS Group | CEA Group
Number analyzed (Participants) | 1089 | 364
percentage of partcipants | 98.4 | 96.7

11. Secondary Outcome: Freedom From Clinically Indicated Target Lesion Revascularization
Description: as for outcome 7
Time Frame: 0 to 1825 days
Measure: Number; unit: percentage of partcipants
Arm/Group | CAS Group | CEA Group
Number analyzed (Participants) | 1089 | 364
percentage of partcipants | 98.4 | 96.7

12. Secondary Outcome: Freedom From Ipsilateral Stroke
Description: Ipsilateral stroke was defined as stroke in the vascular distribution of the study carotid artery. If a subject experienced a bilateral stroke it was counted as an ipsilateral stroke for analysis purposes.
Time Frame: 31 to 365 days
Measure: Number; unit: percentage of participants
Arm/Group | CAS Group | CEA Group
Number analyzed (Participants) | 1049 | 333
percentage of participants | 99.4 | 99.1

13. Secondary Outcome: Freedom From Ipsilateral Stroke
Description: as for outcome 12
Time Frame: 31 to 730 days
Measure: Number; unit: percentage of participants
Arm/Group | CAS Group | CEA Group
Number analyzed (Participants) | 1049 | 333
percentage of participants | 99.0 | 98.7

14. Secondary Outcome: Freedom From Ipsilateral Stroke
Description: as for outcome 12
Time Frame: 31 to 1095 days
Measure: Number; unit: percentage of participants
Arm/Group | CAS Group | CEA Group
Number analyzed (Participants) | 1049 | 333
percentage of participants | 98.4 | 97.8

15. Secondary Outcome: Freedom From Ipsilateral Stroke
Description: as for outcome 12
Time Frame: 31 to 1460 days
Measure: Number; unit: percentage of participants
Arm/Group | CAS Group | CEA Group
Number analyzed (Participants) | 1049 | 333
percentage of participants | 97.8 | 97.3

16. Secondary Outcome: Freedom From Ipsilateral Stroke
Description: as for outcome 12
Time Frame: 31 to 1825 days
Measure: Number; unit: percentage of participants
Arm/Group | CAS Group | CEA Group
Number analyzed (Participants) | 1049 | 333
percentage of participants | 97.8 | 97.3

17. Secondary Outcome: Freedom From Mortality
Time Frame: 0 to 365 days
Measure: Number; unit: percentage of participants
Arm/Group | CAS Group | CEA Group
Number analyzed (Participants) | 1089 | 364
percentage of participants | 98.5 | 99.1

18. Secondary Outcome: Freedom From Mortality
Time Frame: 0 to 730 days
Measure: Number; unit: percentage of participants
Arm/Group | CAS Group | CEA Group
Number analyzed (Participants) | 1089 | 364
percentage of participants | 96.2 | 98.4

19. Secondary Outcome: Freedom From Mortality
Time Frame: 0 to 1095 days
Measure: Number; unit: percentage of partcipants
Arm/Group | CAS Group | CEA Group
Number analyzed (Participants) | 1089 | 364
percentage of partcipants | 94.3 | 97.5

20. Secondary Outcome: Freedom From Mortality
Time Frame: 0 to 1460 days
Measure: Number; unit: percentage of participants
Arm/Group | CAS Group | CEA Group
Number analyzed (Participants) | 1089 | 364
percentage of participants | 91.5 | 93.7

21. Secondary Outcome: Freedom From Mortality
Time Frame: 0 to 1825 days
Measure: Number; unit: percentage of participants
Arm/Group | CAS Group | CEA Group
Number analyzed (Participants) | 1089 | 364
percentage of participants | 87.1 | 89.4

22. Secondary Outcome: Freedom From All Stroke
Time Frame: 0 to 365 days
Measure: Number; unit: percentage of participants
Arm/Group | CAS Group | CEA Group
Number analyzed (Participants) | 1089 | 364
percentage of participants | 96.5 | 97.7

23. Secondary Outcome: Freedom From All Stroke
Time Frame: 0 to 730 days
Measure: Number; unit: percentage of participants
Arm/Group | CAS Group | CEA Group
Number analyzed (Participants) | 1089 | 364
percentage of participants | 95.8 | 96.2

24. Secondary Outcome: Freedom From All Stroke
Time Frame: 0 to 1095 days
Measure: Number; unit: percentage of participants
Arm/Group | CAS Group | CEA Group
Number analyzed (Participants) | 1089 | 364
percentage of participants | 94.5 | 95.3

25. Secondary Outcome: Freedom From All Stroke
Time Frame: 0 to 1460 days
Measure: Number; unit: percentage of participants
Arm/Group | CAS Group | CEA Group
Number analyzed (Participants) | 1089 | 364
percentage of participants | 93.8 | 94.7

26. Secondary Outcome: Freedom From All Stroke
Time Frame: 0 to 1825 days
Measure: Number; unit: percentage of participants
Arm/Group | CAS Group | CEA Group
Number analyzed (Participants) | 1089 | 364
percentage of participants | 93.1 | 94.7

27. Secondary Outcome: Death (Non-Hierarchical)
Time Frame: ≤ 30 Days Post Index Procedure
Population: Analysis population Includes only the most serious event for each subject and includes only each subject's first occurrence of the event. Subjects who did not complete 30 day follow-up and did not have any death, stroke or MI events are excluded.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CAS Group | CEA Group
Number analyzed (Participants) | 1072 | 348
percentage of participants | 0.1 [0.0 to 0.5] | 0.3 [0.0 to 1.6]

28. Secondary Outcome: All Stroke (Non-Hierarchical)
Time Frame: ≤ 30 Days Post Index Procedure
Population: as for outcome 27
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CAS Group | CEA Group
Number analyzed (Participants) | 1072 | 348
percentage of participants | 2.8 [1.9 to 4.0] | 1.4 [0.5 to 3.3]

29. Secondary Outcome: Myocardial Infarction (MI) (Non-Hierarchical)
Time Frame: ≤ 30 Days Post Index Procedure
Population: as for outcome 27
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CAS Group | CEA Group
Number analyzed (Participants) | 1072 | 348
percentage of participants | 0.5 [0.2 to 1.1] | 0.9 [0.2 to 2.5]

30. Secondary Outcome: Death, Stroke or Myocardial Infarction (MI) (Hierarchical)
Time Frame: ≤ 30 Days Post Index Procedure
Population: as for outcome 27
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CAS Group | CEA Group
Number analyzed (Participants) | 1072 | 348
percentage of participants | 3.3 [2.3 to 4.5] | 2.6 [1.2 to 4.9]

31. Secondary Outcome: Death or Stroke (Hierarchical)
Time Frame: ≤ 30 Days Post Index Procedure
Population: as for outcome 27
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CAS Group | CEA Group
Number analyzed (Participants) | 1072 | 348
percentage of participants | 2.9 [2.0 to 4.1] | 1.7 [0.6 to 3.7]

32. Secondary Outcome: Death or Major Stroke (Hierarchical)
Time Frame: ≤ 30 Days Post Index Procedure
Population: as for outcome 27
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CAS Group | CEA Group
Number analyzed (Participants) | 1072 | 348
percentage of participants | 0.6 [0.2 to 1.2] | 0.6 [0.1 to 2.1]

33. Secondary Outcome: Freedom From Death, Stroke and MI Within 30 Days and Ipsilateral Stroke From 31 Days to 5 Years
Time Frame: 0 to 5 years
Measure: Number; unit: percentage of participants
Arm/Group | CAS Group | CEA Group
Number analyzed (Participants) | 1089 | 364
percentage of participants | 94.6 | 94.8

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | CAS Group | CEA Group
Serious Adverse Events (participants affected / at risk) | 376/1089 | 118/364
Other Adverse Events (participants affected / at risk) | 635/1089 | 216/364
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CAS Group (N=1089) | CEA Group (N=364)
Bleeding (Injury, poisoning and procedural complications) | 7 (8) | 3 (3)
Hematoma (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)
Infection (Injury, poisoning and procedural complications) | 3 (6) | 3 (3)
Occlusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vessel trauma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Epistaxis (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
GI bleed (Blood and lymphatic system disorders) | 15 (15) | 8 (8)
Genitourinary (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Vascular (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 13 (15) | 3 (3)
Abnormal lab test (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 22 (25) | 4 (5)
Cardiac arrest (Cardiac disorders) | 5 (5) | 3 (3)
Congestive heart failure (Cardiac disorders) | 10 (12) | 1 (1)
Coronary artery disease (Cardiac disorders) | 57 (70) | 21 (25)
Pulmonary hypertension (Cardiac disorders) | 2 (2) | 0 (0)
Structural heart disease (Cardiac disorders) | 2 (2) | 0 (0)
Myocardial infarction (Cardiac disorders) | 14 (16) | 5 (5)
Hypertension (Vascular disorders) | 6 (6) | 2 (2)
Hypotension (Vascular disorders) | 7 (8) | 1 (1)
Syncope (Vascular disorders) | 4 (4) | 1 (1)
Confusion (Nervous system disorders) | 1 (1) | 0 (0)
Cranial nerve palsy (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 3 (3)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hyperperfusion syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Neurologic other (Nervous system disorders) | 13 (13) | 3 (5)
Peripheral neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 5 (7) | 1 (1)
Subdural hematoma (Nervous system disorders) | 2 (2) | 0 (0)
TIA (Nervous system disorders) | 7 (8) | 2 (2)
Visual disturbance (Nervous system disorders) | 3 (3) | 0 (0)
Ipsilateral major (Nervous system disorders) | 7 (7) | 1 (1)
Ipsilateral minor (Nervous system disorders) | 20 (20) | 6 (6)
Non-ipsilateral major (Nervous system disorders) | 2 (2) | 0 (0)
Non-ipsilateral minor (Nervous system disorders) | 3 (3) | 0 (0)
Anesthesia/Procedural medication related (Surgical and medical procedures) | 0 (0) | 2 (2)
Arrhythmia (Surgical and medical procedures) | 17 (18) | 3 (3)
Bleeding (Surgical and medical procedures) | 11 (11) | 0 (0)
Cranial nerve injury (Surgical and medical procedures) | 2 (2) | 3 (3)
Fluid overload (Surgical and medical procedures) | 1 (1) | 0 (0)
Headache (Surgical and medical procedures) | 0 (0) | 1 (1)
Heparin induced thrombocytopenia (Surgical and medical procedures) | 1 (1) | 0 (0)
Hypertension (Surgical and medical procedures) | 5 (6) | 7 (7)
Hypotension (Surgical and medical procedures) | 69 (69) | 7 (7)
Spasm (Surgical and medical procedures) | 1 (1) | 0 (0)
Urinary retention (Surgical and medical procedures) | 1 (1) | 2 (2)
Vessel trauma (Surgical and medical procedures) | 7 (7) | 0 (0)
Abdominal Aortic Aneurysm (Vascular disorders) | 2 (2) | 2 (2)
Carotid artery disease (Vascular disorders) | 1 (1) | 0 (0)
Contralateral stenosis (Vascular disorders) | 7 (7) | 3 (3)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Occlusion (Vascular disorders) | 1 (1) | 0 (0)
Peripheral vascular disease (Vascular disorders) | 41 (56) | 11 (20)
Pulmonary embolism (Vascular disorders) | 1 (1) | 0 (0)
Renal artery disease (Vascular disorders) | 10 (10) | 1 (1)
Restenosis (Vascular disorders) | 1 (1) | 0 (0)
Stenosis (Vascular disorders) | 3 (3) | 1 (1)
Target lesion restenosis (Vascular disorders) | 8 (8) | 9 (10)
Allergic reaction (Immune system disorders) | 2 (2) | 0 (0)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 21 (23) | 8 (10)
Gastrointestinal (Gastrointestinal disorders) | 29 (39) | 3 (3)
Genitourinary (General disorders) | 25 (28) | 1 (1)
Infection (Infections and infestations) | 23 (25) | 6 (6)
Mental health related (Psychiatric disorders) | 4 (4) | 2 (3)
Metabolic (Metabolism and nutrition disorders) | 10 (10) | 1 (1)
Miscellaneous (General disorders) | 14 (14) | 4 (6)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 41 (45) | 7 (7)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 19 (24) | 9 (9)
Trauma (General disorders) | 13 (15) | 6 (6)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CAS Group (N=1089) | CEA Group (N=364)
Anesthesia/Procedural medication related (Injury, poisoning and procedural complications) | 65 (70) | 51 (55)
Arrhythmia (Injury, poisoning and procedural complications) | 140 (148) | 20 (20)
Cranial nerve injury (Injury, poisoning and procedural complications) | 14 (15) | 48 (51)
Headache (Injury, poisoning and procedural complications) | 73 (74) | 30 (31)
Hypertension (Injury, poisoning and procedural complications) | 40 (40) | 29 (29)
Hypotension (Injury, poisoning and procedural complications) | 252 (268) | 35 (36)
Pain (Injury, poisoning and procedural complications) | 56 (60) | 64 (66)
Other (Gastrointestinal disorders) | 93 (115) | 33 (41)
Other (Infections and infestations) | 81 (92) | 23 (31)
Other (Metabolism and nutrition disorders) | 51 (58) | 24 (25)
Other (General disorders) | 107 (140) | 40 (47)
Other (Musculoskeletal and connective tissue disorders) | 173 (211) | 28 (36)
Other (Respiratory, thoracic and mediastinal disorders) | 56 (66) | 18 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days